CLINICAL TRIAL: NCT03408834
Title: The Effect of Fluid Management by Pleth Variability Index on Acute Kidney Injury in Obese
Brief Title: The Effect of Fluid Management by Pleth Variability Index on Acute Kidney Injury in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Associated professor, Ankara University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-823-16
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Laparoscopic Colorectal Surgery; Acute Kidney Injury
Keywords: NGAL; PVI
MeSH Terms: conditions — Acute Kidney Injury | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulse variability index (Active Comparator): fluid management performed by pulse variability index
  Interventions: Other: pulse variability index
- conventional fluid management (Placebo Comparator): fluid management performed by conventional fluid management
  Interventions: Other: pulse variability index

INTERVENTIONS:
Other: pulse variability index — fluid management with pulse variability index or conventional
  Other Names: conventional

SUMMARY:
This study was to find out whether laparoscopic colorectal surgery is detrimental to the kidneys via PVI monitoring. To detect the kidney injury, so-called kidney troponin NGAL ,which gives earlier information than creatin in renal ischemic injury, was used.

DETAILED DESCRIPTION:
Our object in this study was to find out whether laparoscopic colorectal surgery is detrimental to the kidneys via PVI monitoring. To detect the kidney injury, so-called kidney troponin NGAL ,which gives earlier information than creatine in renal ischemic injury, was used.

Patients undergoing elective laparoscopic colorectal surgery, 18 to 75 years old, planned surgery duration longer than 2 hours, were included in this study. Patients were divided into 2 groups with respect to their fluid resuscitation, Group 1: goal directed fluid therapy via PVI monitoring Group 2: conventional fluid resuscitation. Blood samples were drawn from both groups for NGAL measurement before CO2 insufflation (T0), and at 6th(T1) and 12th(T2) hours after CO2 insufflation. At the end of the surgery, sugammadex was given to all patients for reversal of muscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic surgery
* obese patient

Exclusion Criteria:

* patient refusal
* major comorbidity
* renal failure
* diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2017-09-02 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Diagnosis of acute kidney injury | postoperative 6 th hour
  following up diagnosis of acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIMGUCLU, Study Chair — Ankara University

IPD SHARING:
Plan to Share IPD: No